CLINICAL TRIAL: NCT03702309
Title: Liquid Biopsy Evaluation and Repository Development at Princess Margaret
Acronym: LIBERATE
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: LIBERATE
Record Dates: First submitted 2018-09-25; First posted 2018-10-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Breast Cancer; Lung Cancer; Colon Cancer; Ovarian Cancer; Melanoma; Lymphoma; Leukemia; Mutation; Lynch Syndrome; Cowden Syndrome; BRCA1 Mutation; BRCA2 Mutation; Uterine Cancer; Myeloma; Kidney Cancer; Head and Neck Cancer; Meningioma
Keywords: High Risk; Liquid Biopsy; Circulating Tumor DNA; Blood; Molecular Profiling; Next Generation Sequencing; Solid Tumors; Hematological
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Lung Neoplasms; Colonic Neoplasms; Ovarian Neoplasms; Melanoma; Lymphoma; Leukemia; Colorectal Neoplasms, Hereditary Nonpolyposis; Hamartoma Syndrome, Multiple; Uterine Neoplasms; Neoplasms, Plasma Cell; Kidney Neoplasms; Head and Neck Neoplasms; Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected serially for DNA extraction Archived tissue samples collected for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LIBERATE: Patients with either histological confirmation of a solid tumor or hematological malignancy, or patients identified as high-risk for cancer (based on identified aberration in cancer predisposition gene or on hormonal and/or family history without known aberration).

SUMMARY:
The objective of this protocol is to develop an institution-wide liquid biopsy protocol that will establish a common process for collecting blood and corresponding archived tumor specimens for future research studies at the University Health Network's Princess Margaret Cancer Centre. Circulating cell-free nucleic acids (cfNA), including cell-free DNA (cfDNA) and cell-free RNA (cfRNA), are non-invasive, real-time biomarkers that can provide diagnostic and prognostic information before cancer diagnosis, during cancer treatment, and at disease progression. Cancer research scientists and clinicians at the Princess Margaret are interested in incorporating the collection of peripheral blood samples ("liquid biopsies") into research protocols as a means of non-invasively assessing tumor progression and response to treatment at multiple time points during a patient's course of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with either histological confirmation of a solid tumor or hematological malignancy, OR patients identified as high-risk for cancer (based on identified aberration in cancer predisposition gene or on hormonal and/or family history without known aberration).
2. Patient must be ≥ 18 years old.
3. All patients must have signed and dated an informed consent form for this LIBERATE study.
4. If patients are being co-consented for a separate primary research study listed in Appendix I, they must fulfill the eligibility criteria for that separate primary research study. If there is a discrepancy in the eligibility criteria between protocols, the separate primary research study's criteria take precedence.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors or hematological malignancy and patients identified as high-risk for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-08-03 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Collection and annotation of biospecimens | Through study completion, up to 5 years
  Facilitate and streamline the collection, banking, and annotation of biospecimens (especially liquid biopsy specimens and optionally corresponding archived tumor specimens) for research studies across the University Health Network institution

SECONDARY OUTCOMES:
Electronic Consenting | Through study completion, up to 5 years
  Implement an electronic informed consent process for clinical research at the Princess Margaret Cancer Centre
Correlative Studies Questionnaire | Through study completion, up to 5 years
  Collect observational/epidemiological data using a Correlative Studies Questionnaire for clinical annotation of specimens and future research use. Data collected involves demographics such as family history, medical history, smoking history, and lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Potential to share de-identified study data (including genetic data) with approved research collaborators.

REFERENCES:
- [Derived] Zhao D, Lang N, Liu T, Shelton V, Rangel-Patino J, Gong IY, Hong M, Travas A, Murad V, Alrekhais I, Metser U, Prica A, Kukreti V, Bhella S, Vijenthira A, Crump M, Kuruvilla J, Arruda A, Minden MD, Lam B, Kridel R. Risk Assessment With Ultra-Low-Pass Whole-Genome Sequencing of Cell-Free DNA for Large B-Cell Lymphoma. JCO Precis Oncol. 2025 Jul;9:e2500200. doi: 10.1200/PO-25-00200. Epub 2025 Jul 9. PMID 40632977
- [Derived] Han K, Zou J, Zhao Z, Baskurt Z, Zheng Y, Barnes E, Croke J, Ferguson SE, Fyles A, Gien L, Gladwish A, Lecavalier-Barsoum M, Lheureux S, Lukovic J, Mackay H, Marchand EL, Metser U, Milosevic M, Taggar AS, Bratman SV, Leung E. Clinical Validation of Human Papilloma Virus Circulating Tumor DNA for Early Detection of Residual Disease After Chemoradiation in Cervical Cancer. J Clin Oncol. 2024 Feb 1;42(4):431-440. doi: 10.1200/JCO.23.00954. Epub 2023 Nov 16. PMID 37972346
- [Derived] Sanz-Garcia E, Genta S, Chen X, Ou Q, Araujo DV, Abdul Razak AR, Hansen AR, Spreafico A, Bao H, Wu X, Siu LL, Bedard PL. Tumor-Naive Circulating Tumor DNA as an Early Response Biomarker for Patients Treated With Immunotherapy in Early Phase Clinical Trials. JCO Precis Oncol. 2023 Apr;7:e2200509. doi: 10.1200/PO.22.00509. PMID 37027812
- [Derived] Spiliopoulou P, Janse van Rensburg HJ, Avery L, Kulasingam V, Razak A, Bedard P, Hansen A, Chruscinski A, Wang B, Kulikova M, Chen R, Speers V, Nguyen A, Lee J, Coburn B, Spreafico A, Siu LL. Longitudinal efficacy and toxicity of SARS-CoV-2 vaccination in cancer patients treated with immunotherapy. Cell Death Dis. 2023 Jan 20;14(1):49. doi: 10.1038/s41419-022-05548-4. PMID 36670100
- [Derived] Watson GA, Sanz-Garcia E, Zhang WJ, Liu ZA, Yang SC, Wang B, Liu S, Kubli S, Berman H, Pfister T, Genta S, Spreafico A, Hansen AR, Bedard PL, Lheureux S, Abdul Razak A, Cescon D, Butler MO, Xu W, Mak TW, Siu LL, Chen E. Increase in serum choline levels predicts for improved progression-free survival (PFS) in patients with advanced cancers receiving pembrolizumab. J Immunother Cancer. 2022 Jun;10(6):e004378. doi: 10.1136/jitc-2021-004378. PMID 35705312
- See also: Princess Margaret Cancer Genomics Program — http://www.cancergenomicsprogram.ca/